CLINICAL TRIAL: NCT02835664
Title: Effects of Nicotinamide Riboside on Metabolic Health in (Pre)Obese Humans
Brief Title: Nicotinamide Riboside and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL58119.068.16
Record Dates: First submitted 2016-07-08; First posted 2016-07-18 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Insulin Resistance
Keywords: Nicotinamide Riboside; Obesity; Metabolic health; Insulin resistance; Mitochondrial function; Brown adipose tissue; Energy expenditure; Ectopic lipid accumulation; Cardiovascular risk; Acetylcarnitine
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotinamide Riboside (Experimental): Supplementation of Nicotinamide Riboside (Niagen) of 1000 mg/day for 6 weeks. 2 capsules in the morning together with breakfast and 2 capsules around noon together with lunch. Each capsule contains 250 mg.
  Interventions: Dietary Supplement: Nicotinamide Riboside (Niagen); Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Supplementation of Placebo of 1000 mg/day for 6 weeks. 2 capsules in the morning together with breakfast and 2 capsules around noon together with lunch. Each capsule contains 250 mg.
  Interventions: Dietary Supplement: Nicotinamide Riboside (Niagen); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (Niagen)
Dietary Supplement: Placebo

SUMMARY:
This study will investigate the effects of 6 week Nicotinamide Riboside supplementation (1000 mg/day) on metabolic health in healthy (pre)obese humans. The primary objective will be hepatic and whole body insulin sensitivity. Secondary objectives, to provide information about the underlying mechanism, will be muscle mitochondrial function, brown fat activity, ectopic lipid accumulation, energy metabolism, cardiovascular risk parameters, body composition and acetylcarnitine levels.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian
* Males and postmenopausal females
* Aged 45-65 years at start of the study
* Body mass index (BMI) 27 - 35 kg/m2
* Stable dietary habits (no weight loss or gain >5kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of sports per week)

Exclusion Criteria:

* Type 2 diabetes
* Active diseases (cardiovascular, diabetes, liver, kidney, cancer or other)
* Contra-indication for MRI
* Participation in earlier research or medical examination that included PET/CT scanning
* Alcohol consumption of >2 servings per day
* Smoking in the past 6 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity: muscle- and liver specific | 6 weeks after supplementation
  Hyperinsulinemic euglycemic clamp: Rate of glucose disappearance (Rd) will be calculated by using tracer kinetics.

SECONDARY OUTCOMES:
Muscle mitochondrial function (ex vivo) | 6 weeks after supplementation
  Ex vivo mitochondrial function in skeletal muscle measured by oxygen consumption in muscle fibres (muscle biopsy vastus lateralis) on lipid-derived and carbohydrate-derived substrates.
Ectopic lipid accumulation | 6 weeks after supplementation
  Liver and skeletal muscle lipid accumulation measured with H-MRS in vivo.
Brown adipose tissue activity | 6 weeks after supplementation
  Subjects will be exposed to an individualized cooling protocol, after which an 18F-FDG PET/CT scan is made
Cardiovascular risk parameters | 6 weeks after supplementation
  Cardiac energy status measured with P-MRS and Ambulatory blood pressure.
Whole body energy expenditure | 6 weeks after supplementation
  Sleeping metabolic rate measured during an overnight stay in a respiration chamber.
  Resting metabolic rate measured with ventilated hood system, basal, during insulin stimulation (clamp) and during cold stimulation (cooling protocol BAT activity).
Body composition | 6 weeks after supplementation
  Fat mass and fat free mass measured with a BodPod.
Acetylcarnitine levels | 6 weeks after supplementation
  Skeletal muscle acetylcarnitine levels measured with H-MRS in vivo, before and after exercise stimulation (cycling).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Nascimento EBM, Moonen MPB, Remie CME, Gariani K, Jorgensen JA, Schaart G, Hoeks J, Auwerx J, van Marken Lichtenbelt WD, Schrauwen P. Nicotinamide Riboside Enhances In Vitro Beta-adrenergic Brown Adipose Tissue Activity in Humans. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1437-1447. doi: 10.1210/clinem/dgaa960. PMID 33524145
- [Derived] Remie CME, Roumans KHM, Moonen MPB, Connell NJ, Havekes B, Mevenkamp J, Lindeboom L, de Wit VHW, van de Weijer T, Aarts SABM, Lutgens E, Schomakers BV, Elfrink HL, Zapata-Perez R, Houtkooper RH, Auwerx J, Hoeks J, Schrauwen-Hinderling VB, Phielix E, Schrauwen P. Nicotinamide riboside supplementation alters body composition and skeletal muscle acetylcarnitine concentrations in healthy obese humans. Am J Clin Nutr. 2020 Aug 1;112(2):413-426. doi: 10.1093/ajcn/nqaa072. PMID 32320006